CLINICAL TRIAL: NCT03928925
Title: Bougie or Stylet In Patients Undergoing Intubation Emergently (BOUGIE): a Randomized, Multi-center Trial
Brief Title: Bougie or Stylet In Patients Undergoing Intubation Emergently (BOUGIE)
Acronym: BOUGIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Casey, Research Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 182123
Record Dates: First submitted 2019-04-19; First posted 2019-04-26 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Acute Respiratory Failure
Keywords: Intubation; Bougie

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BOUGIE (Active Comparator): For patients randomized to use of a bougie, the operator will use a bougie on the first attempt at intubation. If successful, an assistant will load an endotracheal tube over the bougie, and the operator (without removing the laryngoscope from the mouth) will guide the tube through the vocal cords to the desired depth in the trachea.
  If the bougie is not successfully placed in the trachea or the endotracheal tube cannot be successfully advanced over the bougie on the first attempt at intubation, the operator may use any approach during subsequent attempts at tracheal intubation.
  Interventions: Other: Bougie
- Endotracheal Tube with Stylet (Active Comparator): For patients randomized to use of an endotracheal tube with stylet, the operator will use an endotracheal tube containing a removeable, malleable stylet, on the first attempt at intubation.
  Manipulation of the shape/curve of the endotracheal tube with stylet is at the discretion of the operator, however a "straight-to-cuff" shape and a bend angle of 25° to 35° is encouraged. The stylet will be left in place until the tube is advanced to the trachea.
  If the endotracheal tube with stylet is not successfully placed in the trachea on the first attempt at intubation, the operator may use any approach during subsequent attempts at tracheal intubation.
  Interventions: Other: Endotracheal Tube with Stylet

INTERVENTIONS:
Other: Bougie — disposable tracheal tube introducer of approximately 70 cm in length
  Arms: BOUGIE
Other: Endotracheal Tube with Stylet — endotracheal tube preloaded with a removable, malleable stylet
  Arms: Endotracheal Tube with Stylet

SUMMARY:
Complications are common during tracheal intubations performed outside of the operating room. Successful intubation on the first attempt has been associated with a lower rate of procedural complications, but the proportion of critically ill patients intubated on the first attempt during tracheal intubations outside of the operating room is less than 90%. The bougie, a thin semi-rigid tube that can be placed into the trachea, allowing a Seldinger-like technique of intubating a patient's airway, has been traditionally reserved for difficult or failed airways. However, a recent single center trial of adult patients intubated in an emergency department demonstrated that use of the bougie on the first attempt improved intubation success, compared to use of a traditional stylet.

Theinvestigators propose a multi-center randomized trial to compare first-attempt bougie use versus endotracheal tube with stylet use for tracheal intubation of critically ill adults in the ED and ICU.

DETAILED DESCRIPTION:
The BOUGIE trial is a prospective, parallel group, pragmatic, randomized trial comparing the effect of bougie use versus endotracheal tube with stylet use on the incidence of successful intubation on the first attempt among adults undergoing urgent or emergent tracheal intubation.

Patients admitted to the study units who are deemed by their clinical team to require intubation and fulfill inclusion criteria without meeting exclusion criteria will be randomized 1:1 to use of a bougie or use of an endotracheal tube and stylet on the first attempt at intubation. All other decisions regarding airway management, including the choice to use a bougie or endotracheal tube and stylet on subsequent attempts, will remain at the discretion of the treating provider.

The trial will enroll 1,106 patients. Conduct of the trial will be overseen by a Data Safety Monitoring Board. An interim analysis will be performed after the enrollment of 553 patients. The analysis of the trial will be conducted in accordance with a pre-specified statistical analysis plan, which will be submitted for publication or made publicly available prior to the conclusion of enrollment.

The primary outcome is successful intubation on the first attempt

The secondary outcome is severe hypoxemia (lowest arterial oxygen saturation between induction and two minutes following intubation of less than 80%)

ELIGIBILITY:
Inclusion Criteria:

1. Patient is located in a participating unit of an adult hospital
2. Planned procedure is tracheal intubation with sedative administration (or tracheal intubation without sedative administration during cardiac arrest)
3. Planned operator is a clinician expected to routinely perform tracheal intubation in the participating unit
4. Planned laryngoscopy device is a non-hyperangulated laryngoscope blade

Exclusion Criteria:

1. Patient is pregnant
2. Patient is a prisoner
3. Urgency of intubation precludes safe performance of study procedures
4. Operator feels an approach to intubation other than use of a bougie or use of an endotracheal tube with stylet would be best for the care of the patient
5. Operator feels use of a bougie is required or contraindicated for the care of the patient
6. Operator feels use of an endotracheal tube with stylet is required or contraindicated for the care of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1106 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Number of intubations with successful intubation on the first attempt | from induction to 2 minutes following tracheal intubation
  The primary outcome is successful intubation on the first attempt. Successful intubation on the first attempt is defined as placement of an endotracheal tube in the trachea (confirmed by standard means including capnography) following: (1) a single insertion of a laryngoscope blade into the mouth and (2) EITHER a single insertion of a bougie into the mouth followed by a single insertion of an endotracheal tube into the mouth OR a single insertion of an endotracheal tube with stylet into the mouth.

SECONDARY OUTCOMES:
Number of intubations with severe hypoxemia | from induction to 2 minutes following tracheal intubation
  Defined as an oxygen saturation less than 80% during the time interval from induction to two minutes after completion of the intubation procedure

OTHER OUTCOMES:
Cormack-Lehane grade of glottic view on first attempt | from induction to 2 minutes following tracheal intubation
  Grade 1: Full view of glottis Grade 2: Partial view of glottis Grade 3: Only epiglottis seen (none of glottis) Grade 4: Neither glottis nor epiglottis seen
Number of laryngoscopy attempts | from induction to 2 minutes following tracheal intubation
Number of attempts at passing bougie | from induction to 2 minutes following tracheal intubation
Number of attempts at passing endotracheal tube | from induction to 2 minutes following tracheal intubation
Duration of intubation | from the first of induction or initiation of laryngoscopy to 2 minutes following tracheal intubation
  The start of the procedure will be defined as either the time of first sedative administration or the time of initiation of laryngoscopy among patients who do not receive a sedative. The end of the procedure will be defined as the time of the final placement of an endotracheal tube within the trachea.
Use of video laryngoscope screen | from induction to 2 minutes following tracheal intubation
  Operator report of use of video laryngoscope screen on first attempt among intubations where the operator used a video laryngoscope
Number of intubations with esophageal intubation | from induction to 2 minutes following tracheal intubation
  Operator report of whether or not an esophageal intubation occurred
Number of intubations with operator-reported aspiration | from induction to 2 minutes following tracheal intubation
  Operator report of whether or not an an aspiration event occurred
Number of intubations with airway trauma | from induction to 2 minutes following tracheal intubation
  Operator report of whether or not airway trauma occurred
Number of intubations with cardiac arrest within 1 hour following intubation | within 1 hour following intubation
Number of intubations with peri-intubation cardiovascular collapse | within 1 hour following intubation
  Defined as any of:
  1. New systolic blood pressure < 65 mmHg between induction and 2 minutes following intubation
  2. New or increased vasopressor between induction and 2 minutes following intubation
  3. Cardiac arrest within 1 hour following intubation
  4. Death within 1 hour following intubation
The number of ICU-free days, for each intubation, in the first 28 days | 28 days
The number of ventilator free days, for each intubation, in the first 28 days | 28 days
The number of patients who experience all-cause in-hospital mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Casey, MD, Study Director — Vanderbilt University Medical Center; Matthew W Semler, MD, MSc, Study Chair — Vanderbilt University Medical Center; Brian E Driver, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis; Matthew E Prekker, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Colorado, Denver, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - University of Iowa Hospital, Iowa City, Iowa
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center | Ochsner Health System, New Orleans, Louisiana
  - Lincoln Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Lexington, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Harborview Medical Center, University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Driver BE, Prekker ME, Klein LR, Reardon RF, Miner JR, Fagerstrom ET, Cleghorn MR, McGill JW, Cole JB. Effect of Use of a Bougie vs Endotracheal Tube and Stylet on First-Attempt Intubation Success Among Patients With Difficult Airways Undergoing Emergency Intubation: A Randomized Clinical Trial. JAMA. 2018 Jun 5;319(21):2179-2189. doi: 10.1001/jama.2018.6496. PMID 29800096
- [Derived] Driver BE, Semler MW, Self WH, Ginde AA, Trent SA, Gandotra S, Smith LM, Page DB, Vonderhaar DJ, West JR, Joffe AM, Mitchell SH, Doerschug KC, Hughes CG, High K, Landsperger JS, Jackson KE, Howell MP, Robison SW, Gaillard JP, Whitson MR, Barnes CM, Latimer AJ, Koppurapu VS, Alvis BD, Russell DW, Gibbs KW, Wang L, Lindsell CJ, Janz DR, Rice TW, Prekker ME, Casey JD; BOUGIE Investigators and the Pragmatic Critical Care Research Group. Effect of Use of a Bougie vs Endotracheal Tube With Stylet on Successful Intubation on the First Attempt Among Critically Ill Patients Undergoing Tracheal Intubation: A Randomized Clinical Trial. JAMA. 2021 Dec 28;326(24):2488-2497. doi: 10.1001/jama.2021.22002. PMID 34879143
- [Derived] Driver B, Semler MW, Self WH, Ginde AA, Gandotra S, Trent SA, Smith LM, Gaillard JP, Page DB, Whitson MR, Vonderhaar DJ, Joffe AM, West JR, Hughes C, Landsperger JS, Howell MP, Russell DW, Gulati S, Bentov I, Mitchell S, Latimer A, Doerschug K, Koppurapu V, Gibbs KW, Wang L, Lindsell CJ, Janz D, Rice TW, Prekker ME, Casey JD; BOUGIE Investigators# and the Pragmatic Critical Care Research Group. BOugie or stylet in patients UnderGoing Intubation Emergently (BOUGIE): protocol and statistical analysis plan for a randomised clinical trial. BMJ Open. 2021 May 25;11(5):e047790. doi: 10.1136/bmjopen-2020-047790. PMID 34035106